CLINICAL TRIAL: NCT04659746
Title: mHealth Technology to Optimize Mental Health in Chronic Patients During the COVID-19 Outbreak in Paraguay
Brief Title: MejoraCare-Paraguay: mHealth Solution for Chronic Patients During the COVID-19 Outbreak in Paraguay
Acronym: MejoraCare_P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Encarnación (Other)
Collaborators: Adhera Health, Inc. (Industry); University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PINV 20-9
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Quality of Life; Stress; Emotional Adjustment
Keywords: COVID-19; Quality of Life; mHealth; Self-efficacy; Emotional Adjustment; Remote Monitoring
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants allocated to the control group will receive the routine care and follow-up for chronic patients in Pandemic situation at Hospital Regional de Encarnación (Encarnación, Paraguay), according to epidemiological surveillance and preventive isolation management protocol released by the Ministry of Health of Paraguay (URL: https://www.mspbs.gov.py/dependencias/portal/adjunto/c1c79a-ProtocoloVigilanciaEpidemiolgica.pdf)
- Intervention (Experimental): Participants allocated to the intervention group will follow the same routine care as the control group. Additionally, they will receive access to the MejoraCare app.
  The MejoraCare app delivers the following functionalities:
  * Remote symptoms monitoring through an electronic Patient Reported Outcome (ePRO)
  * Patient empowerment through personalized educational resources promoting healthy lifestyles
  Interventions: Device: MejoraCare

INTERVENTIONS:
Device: MejoraCare — mHealth solution to support remote monitoring of symptoms and patient empowerment through education.
  Arms: Intervention

SUMMARY:
MejoraCare-Paraguay main objective is to test a mHealth solution (MejoraCare app) to be used for the education and empowerment of chronic patients (COPD, cancer, diabetes, heart disease. hypertension, etc.), and for supporting healthcare professionals to monitor and better understand patients' evolution during the COVID-19 outbreak (MejoraCare dashboard).

This mHealth solution is built upon the Adhera platform, which has already been validated in other therapeutic areas such as smoking cessation.

MejoraCare is expected to raise awareness, educate and empower chronic patients, promoting behavioral changes towards adhering to healthier lifestyles thus reducing the risk of COVID-19 infection while providing emotional regulation support aiming at improving their mental health, quality of life, and emotional well-being.

DETAILED DESCRIPTION:
MejoraCare-Paraguay main objective is to test an mHealth solution (MejoraCare app) to be used for the education and empowerment of chronic patients (COPD, cancer, diabetes, heart disease. hypertension, etc.), and for supporting healthcare professionals to monitor and better understand patients' evolution during the COVID-19 outbreak (MejoraCare dashboard).

This mHealth solution is built upon the Adhera platform, which has already been validated in other therapeutic areas such as smoking cessation.

Its objective is two-fold: on the one hand, MejoraCare will provide the target population with an educational resource to improve their self-efficacy and knowledge about the disease and, on the other hand, to provide them with tools for the regulation of stress, anxiety and negative emotions generated in this high-risk population due to the COVID-19 outbreak situation.

MejoraCare is expected to raise awareness, educate and empower chronic patients, promoting behavioral changes towards adhering to healthier lifestyles thus reducing the risk of COVID-19 infection, while providing emotional regulation support aiming at improving their mental health, quality of life, and emotional well-being.

Personalized health education embedded into MejoraCare app covers the following topics:

* Prevention of COVID-19
* Reinforcement of self-management behaviors for chronic conditions (e.g., physical activity).
* Modules for improving resilience and coping skills related to stress and negative emotions related to the COVID-19 outbreak (e.g., isolation at home).

For health care providers, MejoraCare dashboard provides the following functionalities:

* Segmentation, monitoring, and follow-up of potential positive cases of COVID19 patients and people at special risk
* Support to patients undergoing quarantine at home recovery phase, including remote monitoring of symptoms and a means to contact them in the cases that are deemed necessary by the healthcare professionals.

The specific objectives of MejoraCare-Paraguay are:

1. To analyze the impact of the MejoraCare mHealth solution in terms of mental health, quality of life, and emotional well-being in chronic patients at risk of COVID-19 infection.
2. To analyze the acceptance of the technology by patients and professionals.

This study expects to demonstrate the benefits that an mHealth intervention may have on supporting mental health, quality of life, and emotional well-being for vulnerable patients during the COVID-19 outbreak.

The "info-demia" of constant news about the virus, along with the restrictive/lockdown measures that are being enforced by the governments to reduce the pandemic progression pose a great challenge for the emotional stress for people in general, and with a higher impact on a vulnerable population, especially for those living with chronic conditions that seem to worsen the prognostic in case of infection. Besides, as the pandemic continues its spread, health services are being challenged due to the lack of resources to cope with such a high demand for potential positive cases. In some cases, this affects the quality of care of chronic patients, who also refrain from attending their routine appointments due to the fear of infection. Therefore, reinforcement and behavioral guidance are needed to allow people living with chronic conditions to know and understand which are the measures they need to take to prevent the infection, or how to act in the event that they are infected. Besides, it is necessary to provide this population with tools to support the prevention of psychological and emotional problems that can worsen their health status and, therefore, their quality of life.

mHealth solutions rely on a technology (smartphones) which already has a high level of penetration in the population, makes their widespread highly scalable, and can be released with relatively low costs. If developed under strong quality and safety requirements, they can be a perfect fit for building public health strategies on top of them. On the other hand, the lack of specific digital solutions to educate and empower chronic patients in disease prevention techniques for COVID-19 and other infectious diseases with a relatively high mortality rate among the vulnerable population like the seasonal flu puts them in an even more risky situation to get infected.

ELIGIBILITY:
Inclusion Criteria:

* Legal adults (18+)
* Patients suffering from, at least, one chronic disease.
* Patients owning an Android smartphone and internet connection
* Patients with a minimum level of digital literacy (being able to send text messages)
* Patients able to read and understand Spanish
* Signs the informed consent

Exclusion Criteria:

* Diagnosed with any mental disorder
* Withdraws the consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Change on Health-related Quality of Life | Baseline, 1, and 3, 6 and 12 months
  The Health-related Quality of Life will be measured through the EuroQoL-5D-3L questionnaire measures health related quality of life. The questionnaire consist of five dimensions: mobility, self care, ordinary activities, discomfort, and mood state related to anxiety and depression. Each item ranges form no problem to a lot of problems.

SECONDARY OUTCOMES:
MejoraCare app Usability | 1 month
  Usability of the MejoraCare app will be measured through the SUS questionnaire at the end of the study. This questionnaire will only be completed by patients allocated to intervention group, and gives a global view on the subjective assessment of usability of a technology system
Satisfaction with the MejoraCare app | 1 month
  Satisfaction with the MejoraCare app will be measured through the CSQ questionnaire at the end of the study. This questionnaire will only be completed by patients allocated to the intervention group. This questionnaire is used to measure global patient satisfaction
Change in Self-efficacy | Baseline, 1, 3, 6 and 12 months
  Change in Self-efficacy will be measured through the GSES-12 questionnaire. The scale is composed of 12 items and has 3 factors: Initiative (willingness to initiate behavior), Effort (willingness to make an effort to complete the behavior), and Persistence (persevering to complete the task in the face of adversity).
Change in Anxiety | Baseline, 1, 3, 6 and 12 months
  Change in anxiety will be measured through the GAD-2 questionnaire. The Generalized Anxiety Disorder Questionnaire-2 (GAD-2; Kroenke et al., 2007; García-Campayo et al., 2012) is a 2-item self-report that can be used to screen and detect symptoms of anxiety.
Change in Depression | Baseline, 1, 3, 6 and 12 months
  Change in depression will be measured through the PHQ-2 questionnaire. The Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003; Rodríguez-Muñoz et al., 2017) is a 2-item self-report questionnaire that is used to screen and detect depressive symptomatology. Items responses are rated on a 4-point Likert-scale (0 = not at all, 3 = nearly every day).
Change in Health Empowerment | Baseline, 1, 3, 6 and 12 months
  Change in empowerment will be measured through the EAS questionnaire. The scale measures the degree of empowerment in health-care, assessing self-control, self-efficacy, problem-solving, psychosocial coping, support, motivation, and decision-making
Change in Coping with Stress | Baseline, 1, 3, 6 and 12 months
  Change in coping will be measured through the PSS-4 questionnaire. The short version, PSS-4, is an economical and simple psychological instrument to administer, comprehend, and score. It measures the degree to which situations in one's life over the past month are appraised as stressful.

OTHER OUTCOMES:
Technological profile | Baseline
  It is an ad-hoc scale design to asses the prior knowledge/skill of participants in the use of common technologies as mobiles phones or the computer. The scale has 9 items that score independently in a scale ranging from 0 to 4. Higher scores are associated with a better knowledge in the use of technologies
mHealth App Usability Questionnaire | 1 month
  It is an scale for assess the usability of mHealth applications. The scale has 26 items rated on a 7-point Likert-scale (1 = totally disagree, 7 = totally agree). Higher scores are related to a better opinion regarding the mobile application
Telehealth Questionnaire (TUQ) | 1 month
  It is an scale for assess the utility of mHealth applications. The scale has 16 items rated on a 7-point Likert-scale (1 = totally disagree, 7 = totally agree). Higher scores are related to a better experience regarding the mobile application
COMPUTER FLUENCY SCALE (CFS) | Baseline
  It is a scale to assess the openness of the participant to use technologies in their daily life. The scale has 7 items rated on a 5-point Likert-scale (1 = totally disagree, 5 = totally agree). Higher scores are related to a higher comodity in the use of technologies

CONTACTS AND LOCATIONS:
Overall Officials: Rosa María Baños, PhD, Principal Investigator — Universitat de València-Estudi General
Locations (1):
- Hospital Regional de Encarnación, Encarnación, Itapúa, Paraguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Escriva-Martinez T, Vara MD, Czeraniuk N, Denis M, Nunez-Benjumea FJ, Fernandez-Luque L, Jimenez-Diaz A, Traver V, Llull JJ, Martinez-Millana A, Garces-Ferrer J, Miragall M, Herrero R, Enriquez A, Schaefer V, Cervera-Torres S, Villasanti C, Cabral CV, Fernandez I, Banos RM. mHealth intervention to improve quality of life in patients with chronic diseases during the COVID-19 crisis in Paraguay: A study protocol for a randomized controlled trial. PLoS One. 2022 Nov 8;17(11):e0273290. doi: 10.1371/journal.pone.0273290. eCollection 2022. PMID 36346807